CLINICAL TRIAL: NCT03199430
Title: The Polyphenol Epigallocatechin Gallate Lowers Circulating Catecholamine Concentrations and Alters Lipid Metabolism During Graded Exercise in Man.
Brief Title: Epigallocatechin Gallate Lowers Circulating Catecholamine Concentrations and Alters Lipid Metabolism.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Swansea University (Other)
Responsible Party: Principal Investigator, Liam WIlliams, Postgraduate Student, Swansea University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: PG/2014/28
Record Dates: First submitted 2016-08-03; First posted 2017-06-27 (Actual); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: EGCG Influence on Catecholamine Metabolism
Keywords: catecholamines; Exercise; lipid metabolism
MeSH Terms: conditions — Motor Activity | interventions — epigallocatechin gallate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): 1450mg Corn flour
  Interventions: Dietary Supplement: Placebo
- Epigallocatechin gallate (Active Comparator): 1450mg Epigallocatechin gallate
  Interventions: Dietary Supplement: Epigallocatechin gallate

INTERVENTIONS:
Dietary Supplement: Epigallocatechin gallate
  Arms: Epigallocatechin gallate
Dietary Supplement: Placebo — 1450mg Corn Flour
  Arms: Placebo

SUMMARY:
The aim of this study was to explore the impact of acute ingestion of the polyphenol epigallocatechin galate (EGCG) on catecholamine, catecholamine metabolite, systemic metabolic and cardio-vascular variables across a range of exercise intensities during graded cycle exercise in man.

DETAILED DESCRIPTION:
Written informed consent was obtained from all subjects and all subjects completed the AHA/ACSM health screening questionnaire to ascertain their health status and to show their eligibility to partake in this study.

In a randomized, placebo-controlled, single blind, cross-over design study participants completed two trials after acute consumption of either EGCG or a placebo (PLAC) supplement after an overnight fast. After a two-hour monitoring period following ingestion participants performed a continuous graded cycle exercise test to volitional exhaustion. There was at least a 7-day washout period between trials.

Participants were randomly assigned to either the intervention or placebo trial. After an overnight fast participants arrived to the laboratory and were observed ingesting two capsules each of EGCG (minimum 94% EGCG <0.1% caffeine) from a commercially available brand (TEAVIGO™; TAIYO GmbH, 1450 mg) or a placebo (1450 mg Corn Flour). Capsules were weighed and sorted to within ±5%. The supplement was consumed in two size 00 vegetarian gelatin capsules alongside a standardized amount of distilled water (200ml).

Experimental Protocol Prior to participation in the experimental trials participants were familiarized with the laboratory equipment and the test procedures. On the morning of the test participants reported to the Exercise Physiology Laboratory following an 8-10 hour fast where standard measures of the participants' body mass, (weighting scales; Seca 770 Digital Scales, Seca Ltd, Birmingham, UK) height (stadiometer; Holtain Stadiometer, Holtain Ltd, Cymrych, Wales) and body fat percentage using bioelectrical impedance analysis (Bodystat Quadscan 4000, Bodystat Ltd, Isle of Man, UK) whilst wearing minimal clothing, were taken.

Participants were then seated for a 10-minute period while a cannula was inserted into an antecubital vein. This was connected to a three-way stopcock for the repeated collection of venous blood at rest and during the exercise test. Saline (2-3 ml) was infused regularly keep the cannula patent. After a 10-minute rest period a venous blood sample (7 ml) was collected into a lithium-heparinised vacutainer. In addition, baseline measures of heart rate (Polar RS800CX), and a 10-minute sample of respiratory gas (Jaeger Vyuntus CPX, Erich Jaeger GmbH,CareFusion Hoechbegh, Germany) were also taken at this time. Expired air was measured for the fractional concentration of oxygen (FEO2%) and carbon dioxide (FECO2%) and for the volume of air (SentrySuite Software, Erich Jaeger GmbH,CareFusion Hoechbegh, Germany) expired during the period to allow for determination of volumes of O2 utilization and CO2 production. These data were used for determination of oxidative energy expenditure using principles of indirect calorimetry (Frayn 1983; Jeukendrup & Wallis, 2005).

Following collection of resting parameters participants were rested in a semi-reclined position for two hours. Thereafter, after a 5-minute transition period, participants mounted a cycle ergometer (Lode Excalibur Sport Ergometer, Lode BV Groningen, The Netherlands) to perform a graded exercise test. Participants were instructed to cycle between 60-70 rpm at an initial power output of 60 Watts (W) with an increase in 30 W every 3 minutes. Verbal encouragement was provided to the participant throughout. Heart rate was measured constantly throughout the exercise test in real-time via a telemetry chest strap and wireless receiver (Polar RS800CX) alongside respiratory gas measurements. Two and a half minutes into each stage, a rating of perceived exertion (RPE) was taken from the participant (Borg, 1982) and a venous blood sample taken. The test continued until volitional exhaustion which was defined by the following criteria 1) cadence dropping below 50 rpm, 2) heart rate within 10 beats of age-predicted maximum, 3) levelling off of VO2 though workload had increased. At this point cardio-respiratory variables were recorded and a final blood sample was taken at exhaustion.

Participants were given a food and physical activity diaries to complete in the 72 hours prior to the first experimental trial. Participants were also instructed to avoid alcohol, foods with high polyphenols content and additional green tea consumption during this period. Participants were also instructed not to perform any physical activity in the 24h period immediately prior to the exercise trial.

Blood Analyses Venous blood samples were analysed immediately for lactate and glucose levels (Biosen C-Line, EKF Diagnostics). Thereafter, the remainder of the sample was centrifuged (Heraeus Megafuge 8, Thermo Scientific) for 10 minutes at 3,000 rpm) with ~3ml of plasma extracted into individual 1ml microcentrifuge tubes and frozen immediately (-80°C) for later analysis of metanephrine, normetanephrine and catecholamine (adrenaline and noradrenaline) concentrations using commercially available enzyme linked absorbent assays (ELISA, Eagle Biosciences Inc, Nashua, New Hampshire, USA). Blood points selected for use with the assay kits were, baseline (REST), two hours post ingestion at rest (POST-ING) and during exercise at highest lipid oxidation rate (FATpeak), lactate threshold (LT) and at peak rate of oxygen consumption (VO2peak) for each individual were analysed. Lactate threshold was calculated using Lactate-E software (Newell et al, 2007).

The data was analysed using the Statistical Package for the Social Sciences software (Version 22, SPSS, inc). Data was reported as means±SD with P0.05 accepted. All variables were examined using paired t-tests for comparison of experimental trial differences.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-35 years old. Caffeine intake ≤400 mg.d-1 (thus less than four cups of tea/ coffee or caffeinated soda beverages).

Habitual participation in exercise three to five times per week for 30-90 minutes per formal exercise session.

Exclusion Criteria:

* Female Any injury, assessed via health screening questionnaire prior to the start of the study.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2015-09; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
change in Adrenaline & Noradrenaline concentrations (nmol.l-1) | Relativised to each metabolic domain; rest, 2 hours post ingestion, highest lipid oxidation rate during exercise, lactate threshold and VO2peak (participant dependant)
  Changes in Adrenaline & Noradrenaline concentrations (nmol.l-1) from rest to exhaustion under EGCG and placebo conditions.
Changes in Metanephrine and Normetanephrine (pmol.l-1) | Relativised to each metabolic domain; rest, 2 hours post ingestion, highest lipid oxidation rate during exercise, lactate threshold and VO2peak (participant dependant)
  Changes in Metanephrine & Normetanephrine concentrations (pmol.l-1) from rest to exhaustion under EGCG and placebo conditions.
Changes in lipid and carbohydrate oxidation (g.min-1) | Over a period of approximately 2 and a half hours with the data collected relativised to each metabolic domain; rest, highest lipid oxidation rate during exercise, lactate threshold and VO2peak (participant dependant)
  Changes in lipid and carbohydrate oxidation (g.min-1) from rest to exhaustion under EGCG and placebo conditions.

SECONDARY OUTCOMES:
Changes in blood glucose concentrations (mmol.l-1) | Relativised to each metabolic domain; rest, two hours post ingestion, highest lipid oxidation rate during exercise, lactate threshold and VO2peak (participant dependant)
  Changes in glucose concentrations (pmol.l-1) from rest to exhaustion under EGCG and placebo conditions.
Changes in exercise performance (S) under EGCG and placebo conditions. | over a period of approximately 30 minutes from rest to volitional exhaustion.
  Changes in markers of exercise performance, (performance time) under EGCG and placebo conditions
Changes in blood lactate concentrations (mmol.l-1) | Relativised to each metabolic domain; rest, two hours post ingestion, highest lipid oxidation rate during exercise, lactate threshold and VO2peak (participant dependant)
  Changes in lactate concentrations (pmol.l-1) from rest to exhaustion under EGCG and placebo conditions.
Changes in exercise performance (W) under EGCG and placebo conditions. | over a period of approximately 30 minutes from rest to volitional exhaustion.
  Changes in markers of exercise performance, (maximal power obtained) under EGCG and placebo conditions

REFERENCES:
- [Background] Newell J, Higgins D, Madden N, Cruickshank J, Einbeck J, McMillan K, McDonald R. Software for calculating blood lactate endurance markers. J Sports Sci. 2007 Oct;25(12):1403-9. doi: 10.1080/02640410601128922. PMID 17786693
- [Background] Frayn KN. Calculation of substrate oxidation rates in vivo from gaseous exchange. J Appl Physiol Respir Environ Exerc Physiol. 1983 Aug;55(2):628-34. doi: 10.1152/jappl.1983.55.2.628. PMID 6618956
- [Background] Jeukendrup AE, Wallis GA. Measurement of substrate oxidation during exercise by means of gas exchange measurements. Int J Sports Med. 2005 Feb;26 Suppl 1:S28-37. doi: 10.1055/s-2004-830512. PMID 15702454